CLINICAL TRIAL: NCT04523311
Title: An Evaluation of Brief Online Hypnosis for Migraine and Tension-type Headaches
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Canterbury Christ Church University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PaulDavies2020
Record Dates: First submitted 2020-08-19; First posted 2020-08-21 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Migraine; Tension-Type Headache
MeSH Terms: conditions — Migraine Disorders; Tension-Type Headache | interventions — Hypnosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypnosis + usual care (Experimental): An online, group-based, single session hypnosis workshop followed by 2 weeks of self hypnosis. Participants will continue with whatever usual care they receive/undertake.
  Interventions: Behavioral: Hypnosis.; Other: Usual care
- Waitlist control + usual care (Other): The control group will receive no intervention beyond whatever usual care they receive/undertake. After the study is complete, they will be offered the option of participating in the hypnosis intervention.
  Interventions: Other: Usual care

INTERVENTIONS:
Behavioral: Hypnosis. — Online, group-based, single session hypnosis workshop followed by 2 weeks of self hypnosis.
  Arms: Hypnosis + usual care
Other: Usual care — Participants will be asked to continue with whatever interventions they are already receiving/employing to manage their migraine and tension-type headaches.

SUMMARY:
This study aims to conduct an initial evaluation of whether a single, online, group-based session of hypnosis followed by self-hypnosis can decrease symptoms of migraine and tension-type headaches as well as improve quality of life and perceived self-efficacy over the condition.

DETAILED DESCRIPTION:
This study is a pilot randomised controlled trial (RCT) comparing a single, online, group-based session of hypnosis followed by self-hypnosis for people with migraines or tension-type headaches with a wait-list control. A battery of self-report measures and a 2-week headache diary will be administered online at baseline (weeks 0 and 1), post-intervention (weeks 7 and 8) and at follow-up (weeks 11 and 12).

ELIGIBILITY:
Inclusion Criteria:

* Self-reported diagnosis of migraine or tension-type headaches from a General Practitioner (i.e. family physician) and/or specialist physician.
* Score above the cut-off for either migraine or tension-type headache on the Headache Screening Questionnaire.
* Have experienced at least one headache every two weeks over the last 3 months.
* Otherwise healthy physically and mentally.
* Able to understand written and spoken English.
* Have the IT equipment necessary to access Zoom videoconferencing and the Qualtrics survey system.

Exclusion Criteria:

* Substantial medical or psychiatric co-morbidities including diagnoses of epilepsy, psychosis or personality disorder, and/or taking psychiatric medication.
* A diagnosis of medication overuse headache.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2020-10-27 (Actual); Primary Completion 2021-02-24 (Actual); Study Completion 2021-02-24 (Actual)

PRIMARY OUTCOMES:
Change from baseline at 7-8 weeks in mean headache rating averaged over 2 weeks of headache diary entries. | Post intervention (weeks 7-8)
  At baseline (weeks 0-1) and post-intervention (weeks 7-8), participants will complete a headache diary for two weeks. The diary comprises hourly ratings of headache intensity (during waking hours) on a 0-5 scale, with higher scores indicating greater migraine/tension-type headache symptom burden. The mean rating over two weeks is used.

SECONDARY OUTCOMES:
Change from baseline at 11-12 weeks in mean headache rating averaged over 2 weeks of headache diary entries. | Follow-up (weeks 11-12)
  As described in the primary outcome.
Change from baseline at 7-8 weeks in headache frequency over 2 weeks of headache diary entries. | Post intervention (weeks 7-8)
  Using the aforementioned headache diary, the frequency of headaches over the 2 week diary period will be calculated.
Change from baseline at 11-12 weeks in headache frequency over 2 weeks of headache diary entries. | Follow-up (weeks 11-12)
  Using the aforementioned headache diary, the frequency of headaches over the 2 week diary period will be calculated.
Change from baseline at 7-8 weeks in mean headache duration over 2 weeks of headache diary entries. | Post intervention (weeks 7-8)
  Using the aforementioned headache diary, the mean duration of headaches over the 2 week diary period will be calculated.
Change from baseline at 11-12 weeks in mean headache duration over 2 weeks of headache diary entries. | Follow-up (weeks 11-12)
  Using the aforementioned headache diary, the mean duration of headaches over the 2 week diary period will be calculated.
Change from baseline at week 7 on the Depression, Anxiety and Stress Scales - 21 item version (DASS-21) | Post intervention (week 7)
  This measures symptoms of depression, anxiety and stress producing a score between 0 and 63, with higher scores indicating greater symptomatology.
Change from baseline at week 11 on the Depression, Anxiety and Stress Scales - 21 item version (DASS-21) | Follow-up (week 11)
  This measures symptoms of depression, anxiety and stress producing a score between 0 and 63, with higher scores indicating greater symptomatology.
Change from baseline at week 7 on the Warwick-Edinburgh Mental Wellbeing (WEMWBS) Scale | Post intervention (week 7)
  This measures psychological wellbeing, producing a score between 15 and 75, with higher scores indicating greater wellbeing.
Change from baseline at week 11 on the Warwick-Edinburgh Mental Wellbeing (WEMWBS) Scale | Follow-up (week 11)
  This measures psychological wellbeing, producing a score between 15 and 75, with higher scores indicating greater wellbeing.
Change from baseline at week 7 on the Headache-Specific Locus of Control Scale (HSLC). | Post intervention (week 7)
  This measures one's sense of locus of control over headaches, producing a score between 33 and 165, with higher scores indicating more external perceived locus of control.
Change from baseline at week 11 on the Headache-Specific Locus of Control Scale (HSLC). | Follow-up (week 11)
  This measures one's sense of locus of control over headaches, producing a score between 33 and 165, with higher scores indicating more external perceived locus of control.
Change from baseline at week 7 on the Headache Management Self-efficacy Scale (HMSE). | Post intervention (week 7)
  This measures headache management self-efficacy, producing a score between 25 and 175, with higher scores indicating greater perceived self-efficacy over headache self-management.
Change from baseline at week 11 on the Headache Management Self-efficacy Scale (HMSE). | Follow-up (week 11)
  This measures headache management self-efficacy, producing a score between 25 and 175, with higher scores indicating greater perceived self-efficacy over headache self-management.
Change from baseline at 7-8 weeks in headache related medication consumption over a two week period. | Post intervention (weeks 7-8)
  At baseline (weeks 0-1) and post-intervention (weeks 7-8), participants will keep a diary of their daily, headache-related medication consumption over a two week period. From this, changes in type, dose and frequency of medication will be calculated.
Change from baseline at 11-12 weeks in headache related medication consumption over a two week period. | Follow-up (weeks 11-12)
  At baseline (weeks 0-1) and follow-up (weeks 11-12), participants will keep a diary of their daily, headache-related medication consumption over a two week period. From this, changes in type, dose and frequency of medication will be calculated.

OTHER OUTCOMES:
Baseline scores on the Credibility/Expectancy of Change Questionnaire will moderate the primary and secondary outcomes. | Baseline (week 0)
  This questionnaire measures how much people believe the therapy will help improve lifestyle and functioning prior to the start of the therapy, producing a score between 0 and 21, with higher scores indicating greater treatment credibility and expectancy for change.
Baseline scores on the Attitudes Towards Hypnosis scale will moderate the primary and secondary outcomes specified above. | Baseline (week 0)
  This scale measures how much people believe hypnosis can be helpful, producing a score between 13 and 91, with higher scores indicating greater belief in the efficacy of hypnosis.
Week 2 scores of a bespoke measure of hypnotic suggestibility will predict the degree of change in the primary and secondary outcomes specified above [this applies to the intervention group only]. | Within the online, group-based intervention session (week 2).
  This bespoke measure will be administered in the online, group-based hypnosis session and will measure intervention participants' suggestibility, producing a score from 0 to 50, with higher scores indicating greater suggestibility.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Davies, MSc, Principal Investigator — Canterbury Christ Church University; Fergal Jones, PhD, PsychD, Study Director — Canterbury Christ Church University; Robert Agnew, DClinPsych, Study Director — Private Practice
Locations (1):
- Salomons Institute for Applied Psychology, Royal Tunbridge Wells, United Kingdom